CLINICAL TRIAL: NCT00468845
Title: A Multiple Dose, Randomized, Double-Blind Multicenter Study Of The Efficacy And Safety Of Pregabalin Compared To Placebo In The Treatment Of Patients With Post-Surgical Pain From Hysterectomy
Brief Title: Study Of The Efficacy And Safety Of Pregabalin Compared To Placebo For Treatment Of Post-Surgical Pain From Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081153
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2011-06

CONDITIONS: Pain, Postoperative
Keywords: pain after hysterectomy; amount of opioids used
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: pregabalin (Lyrica)
- 2 (Experimental)
  Interventions: Drug: pregabalin (Lyrica)
- 3 (Placebo Comparator)
  Interventions: Drug: matched placebo

INTERVENTIONS:
Drug: pregabalin (Lyrica) — 150 mg/day double blind (divided doses)
  Arms: 1
Drug: pregabalin (Lyrica) — 300 mg/day double blind (divided doses)
  Arms: 2
Drug: matched placebo — matched placebo
  Arms: 3

SUMMARY:
To assess the efficacy of pregabalin compared to placebo on pain following hysterectomy , measured using subject reported assessments of pain.

ELIGIBILITY:
Inclusion Criteria:

* The subject will have elective total abdominal hysterectomy using a transverse incision with or without bilateral salpingo-oophorectomy. The total hysterectomy may, however, be cervix-sparing.
* The subject is expected to remain at the hospital (or intermediate care facility) for a minimum of 2 days following surgery.
* The subject's preoperative health is graded as the American Society of Anesthesiologist P1 to P2.

Exclusion Criteria:

* Subjects having vaginal hysterectomy (whether laparoscopically assisted or not)
* Subjects having additional procedures (such as those involving the bladder) at the same time as the total abdominal hysterectomy
* The use of nerve block, spinal anesthesia or epidural anesthesia for post-surgical pain control
* Subjects who have been using any opioid medications 2 weeks or more continuously within 3 months prior to the screening visit.
* The subject has taken any NSAID or any analgesic other than acetaminophen within 3 days prior to surgery or is unwilling to abstain from NSAIDs or other analgesics, except as specified in the protocol, during the study. (Subjects taking <325 mg per day of aspirin at a stable dose for at least 30 days before the first dose of study medication will be allowed to continue their aspirin regimen for the duration of the study).

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (9):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
- Canada (3):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site, Prague, Czechia
- Hong Kong (2):
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin
- South Africa (7):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Krugersdorp, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Ladysmith, KwaZulu-Natal
  - Pfizer Investigational Site, Newcastle, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town, Western Cape
  - Pfizer Investigational Site, Parktown
- Spain (3):
  - Pfizer Investigational Site, Cadiz
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Valencia
- Sweden (3):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Stockholm
- Thailand (3):
  - Pfizer Investigational Site, Bangkoknoi, Bangkok
  - Pfizer Investigational Site, Muang, Changwat Khon Kaen
  - Pfizer Investigational Site, Muang, Chiang Mai
- United Kingdom (5):
  - Pfizer Investigational Site, Leicester, Leicestershire
  - Pfizer Investigational Site, Edinburgh, Scotland
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Livingstone

REFERENCES:
- [Derived] Singla NK, Chelly JE, Lionberger DR, Gimbel J, Sanin L, Sporn J, Yang R, Cheung R, Knapp L, Parsons B. Pregabalin for the treatment of postoperative pain: results from three controlled trials using different surgical models. J Pain Res. 2014 Dec 23;8:9-20. doi: 10.2147/JPR.S67841. eCollection 2015. PMID 25565885
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081153&StudyName=Study%20Of%20The%20Efficacy%20And%20Safety%20Of%20Pregabalin%20Compared%20To%20Placebo%20For%20Treatment%20Of%20Post-Surgical%20Pain%20From%20Hysterectomy

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin 150mg: Pregabalin 75 mg twice a day (150 mg/day total)
- Pregabalin 300 mg: Pregabalin 150 mg twice a day (300 mg/day total)
- Placebo: Matching placebo capsule
Period: Overall Study
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Started | 162 | 170 | 169
Received Treatment | 161 | 166 | 167
Completed | 141 | 136 | 139
Not Completed | 21 | 34 | 30
Not completed — Adverse Event | 9 | 14 | 11
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Other | 4 | 9 | 5
Not completed — No longer willing to participate | 5 | 6 | 10
Not completed — Randomized, not treated | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo | Total
Number analyzed (Participants) | 162 | 170 | 169 | 501
Age, Customized [Number; unit: participants]
  25-44 years | 77 | 76 | 88 | 241
  45-70 years | 84 | 90 | 79 | 253
  Unspecified | 1 | 4 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 170 | 169 | 501
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Worst Pain Using the Modified Brief Pain Inventory - Short Form (m-BPI-sf)
Description: Modified Brief Pain Inventory - Short Form (m-BPI-sf): participant rated 11-point Likert rating scale ranged from 0 (no pain) to 10 (worst pain imaginable).
  Least Square (LS) Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Day 2 (24 hours post surgery [PS])
Population: Modified intent-to-treat (mITT) population: participants who received at least 1 dose study drug, had at least 1 post baseline safety and efficacy evaluation, took all pre-surgery medication, had no complications during surgery with discontinuation, no PS infection with additional hospitalization/readmission, had primary efficacy measurement PS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 151 | 149 | 156
Units on a scale | 7.1 (0.18) | 7.2 (0.18) | 7.4 (0.18)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Test type: Superiority or Other; p = 0.1378, ANOVA — Weighted Z-score test method of Fisher (1998) and Cui et al (1999)applied to maintain alpha level. A step down procedure for multiple comparisons to control the maximum experiment wise type I error rate at 0.05 level. 300mg tested prior to 150mg
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Test type: Superiority or Other; p = 0.4710, ANOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Current Pain - Pain With Movement Caused by Sitting
Description: Participant sat upright from supine position, followed by 120 second (sec) rest period, during which participant asked to rate pain with movement. Assessment performed 3 times each day of hospital stay, with 1 daily assessment at 24 (+/- 2) hour interval from end of surgery. Current pain reported on 11 point Likert scale 0 (no pain) to 10 (worst pain imaginable). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Day 1 (day of surgery), up to 7 days PS, Discharge, 2 and 4 weeks PS
Population: mITT; n = number of evaluable participants analyzed for the given time point; N=number of evaluable participants analyzed; Results presented for only those timepoints PS where at least 4 participants in each treatment arm completed the questionnaire at baseline and respective time point.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 147 | 141 | 149
Units on a scale
  24 Hours PS (n=147, 141, 149) | 5.21 (0.188) | 5.53 (0.194) | 5.28 (0.189)
  48 Hours PS (n=142, 141, 142) | 3.57 (0.185) | 3.71 (0.189) | 3.67 (0.189)
  72 Hours PS (n=83, 90, 75) | 2.80 (0.239) | 3.04 (0.225) | 3.20 (0.257)
  96 Hours PS (n=29, 31, 26) | 2.31 (0.425) | 3.20 (0.383) | 3.20 (0.444)
  120 Hours PS (n=14, 15, 12) | 2.89 (0.584) | 2.84 (0.527) | 2.36 (0.633)
  144 Hours PS (n=2, 5, 5) | 1.86 (1.496) | 1.26 (1.177) | 2.00 (1.010)
  Discharge (n=141, 135, 144) | 2.67 (0.175) | 2.99 (0.181) | 2.42 (0.176)
  Day 14 (n=126, 120, 128) | 1.08 (0.140) | 1.37 (0.145) | 1.30 (0.143)
  Day 28 (n=138, 138, 142) | 0.70 (0.126) | 0.91 (0.129) | 0.76 (0.127)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.7752, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.3375, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.7029, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.8618, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.2117, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.6255, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; 96 hours PS; Test type: Superiority or Other; p = 0.0942, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; 96 hours PS; Test type: Superiority or Other; p = 0.9907, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; 120 hours PS; Test type: Superiority or Other; p = 0.4678, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; 120 hours PS; Test type: Superiority or Other; p = 0.5500, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; 144 hours PS; Test type: Superiority or Other; p = 0.9333, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; 144 hours PS; Test type: Superiority or Other; p = 0.7396, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2932, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0164, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.2468, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.7022, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 17: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.7257, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.3854, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

3. Secondary Outcome: Current Pain - Pain With Movement Caused by Peak Expiratory (PEF) Test
Description: Current pain with movement caused by peak expiratory flow (PEF) test as reported by participant on 11 point Likert scale 0 (no pain) to 10 (worst pain). Assessment performed 3 times each day of hospital stay, with 1 daily assessment at 24 (+/- 2) hour interval from end of surgery. PEF test performed 3 times, with 120sec rest periods in between. At beginning of each rest period, participant asked to rate pain caused by forced expiration. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Day 1, up to 7 days PS, 2 and 4 weeks PS
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 146 | 143 | 148
Units on a scale
  24 hours PS (n=146, 142, 148) | 4.83 (0.202) | 4.92 (0.209) | 4.97 (0.207)
  48 hours PS (n=141, 143, 140) | 3.22 (0.204) | 3.47 (0.205) | 3.46 (0.210)
  72 hours PS (n=83, 90, 74) | 2.62 (0.242) | 2.69 (0.228) | 3.04 (0.263)
  96 hours PS (n=28, 31, 25) | 1.88 (0.465) | 3.05 (0.414) | 3.28 (0.487)
  120 hours PS (n=13, 14, 11) | 1.97 (0.685) | 2.10 (0.609) | 1.45 (0.740)
  144 hours PS (n=2, 5, 3) | 3.67 (2.472) | 0.67 (1.453) | 1.67 (1.764)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.5997, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.8582, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.3704, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.9747, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.2033, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.2752, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; 96 hours PS; Test type: Superiority or Other; p = 0.0183, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; 96 hours PS; Test type: Superiority or Other; p = 0.6906, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; 120 hours PS; Test type: Superiority or Other; p = 0.5446, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; 120 hours PS; Test type: Superiority or Other; p = 0.4852, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; 144 hours PS; Test type: Superiority or Other; p = 0.5879, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; 144 hours PS; Test type: Superiority or Other; p = 0.7699, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

4. Secondary Outcome: Area Under the Curve (AUC) Pain - Pain With Movement Caused by Sitting
Description: Time-normalized AUC of pain with movement caused by sitting reported by participants. Participant sat upright from supine position, followed by a 120sec rest period, during which the participant asked to rate pain with movement. Assessment performed 3 times each day of hospital stay, with 1 daily assessment at 24 (+/- 2) hour interval from end of surgery. Current pain reported on 11 point Likert scale 0 (no pain) to 10 (worst pain imaginable). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: 48 +/- 4 hours PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 147 | 140 | 150
Units on a scale | 4.87 (0.155) | 5.01 (0.161) | 4.87 (0.157)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Test type: Superiority or Other; p = 0.9676, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Test type: Superiority or Other; p = 0.4944, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

5. Secondary Outcome: Area Under the Curve (AUC) Pain - Pain With Movement Caused by Peak Expiratory Flow (PEF) Test
Description: Time-normalized AUC of pain reported by participants with movement caused by PEF test. Pain reported by participant on 11 point Likert scale 0 (no pain) to 10 (worst pain). PEF test performed 3 times, with 120sec rest periods in between. At beginning of each rest period, participant asked to rate pain caused by forced expiration. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: 48 +/- 4 hours PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 148 | 142 | 146
Units on a scale | 4.45 (0.167) | 4.64 (0.174) | 4.61 (0.173)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Test type: Superiority or Other; p = 0.4801, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Test type: Superiority or Other; p = 0.8832, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

6. Secondary Outcome: Current Pain at Rest
Description: Pain reported by participants at rest (numeric rating scale (NRS) - Current Pain) on an 11 point Likert scale 0 (no pain) - 10 (worst pain). Pain at rest during the hospital stay was assessed just before each Pain with Movement assessment. Assessment performed 3 times each day of hospital stay, with 1 of daily assessments at 24 (+/- 2 ) hour intervals from end of surgery. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: 8, 16, 24, 32, 40, 48 hours PS
Population: mITT; n = number of evaluable participants analyzed for the given time point; N=number of evaluable participants analyzed
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 151 | 147 | 154
Units on a scale
  8 Hours PS (n=123, 125, 126) | 5.13 (0.232) | 5.39 (0.231) | 5.47 (0.225)
  16 Hours PS (n=94, 88, 107) | 4.06 (0.256) | 4.55 (0.273) | 4.30 (0.245)
  24 Hours PS (n=151, 147, 154) | 3.79 (0.179) | 3.76 (0.184) | 3.93 (0.180)
  32 Hours PS (n=127, 127, 136) | 3.37 (0.207) | 3.31 (0.212) | 3.55 (0.204)
  40 Hours PS (n=93, 97, 100) | 2.97 (0.265) | 2.71 (0.265) | 2.98 (0.263)
  48 Hours PS (n=142, 143, 140) | 2.60 (0.173) | 2.26 (0.174) | 2.65 (0.179)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 8 Hours PS; Test type: Superiority or Other; p = 0.2125, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 8 Hour PS; Test type: Superiority or Other; p = 0.7602, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 16 Hours PS; Test type: Superiority or Other; p = 0.4053, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 16 Hours PS; Test type: Superiority or Other; p = 0.4147, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 24 Hours PS; Test type: Superiority or Other; p = 0.5556, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 24 Hours PS; Test type: Superiority or Other; p = 0.4820, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; 32 Hours PS; Test type: Superiority or Other; p = 0.5088, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; 32 Hours PS; Test type: Superiority or Other; p = 0.3900, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; 40 Hours PS; Test type: Superiority or Other; p = 0.9659, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; 40 Hours PS; Test type: Superiority or Other; p = 0.3968, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; 48 Hours PS; Test type: Superiority or Other; p = 0.8308, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; 48 Hours PS; Test type: Superiority or Other; p = 0.0902, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

7. Secondary Outcome: Area Under the Curve (AUC) of Pain at Rest During the First Two Days of Hospital Stay
Description: Time-normalized AUC of pain reported by participants on 11 point Likert scale 0 (no pain) to 10 (worst pain). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: 48 +/- 4 hours PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 151 | 147 | 154
Units on a scale | 3.62 (0.143) | 3.58 (0.147) | 3.76 (0.144)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Test type: Superiority or Other; p = 0.4388, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Test type: Superiority or Other; p = 0.3364, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

8. Secondary Outcome: Total Cumulative Dose of Opioids Following Surgery
Description: Total cumulative dose was calculated as milligram (mg) of morphine equivalent and included opioids administered by any route. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: 24, 48 Hours PS, Discharge (day 3 up to day 7 PS)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: milligram (mg)
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 150 | 147 | 153
milligram (mg)
  24 hours PS (n=150, 147, 153) | 113.38 (7.078) | 111.27 (7.211) | 124.44 (7.160)
  48 hours PS (n=150, 147, 151) | 148.67 (9.218) | 144.95 (9.391) | 168.31 (9.372)
  Till Discharge (n=147, 143, 144) | 164.28 (11.161) | 167.01 (11.410) | 195.32 (11.569)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.2409, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.1654, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.1110, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.0598, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Till Discharge; Test type: Superiority or Other; p = 0.0398, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Till Discharge; Test type: Superiority or Other; p = 0.0623, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

9. Secondary Outcome: Integrated Analgesic Score
Description: The integrated analgesic score (a combination of opioid use and either worst pain, or pain at rest, or pain caused by sitting, or pain caused by forced expiration as defined by Silverman et al 1993) was the sum of percent differences from mean rank for pain and opioids and ranged from -200 to 200 where lower values represent improvement. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: 0-24, 24-48, 48-72 hours PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 150 | 145 | 151
Units on a scale
  0-24 Hours PS (n=150, 145, 151) | -6.58 (6.795) | -11.66 (6.991) | 3.36 (6.906)
  24-48 Hours PS (n=141, 142, 139) | -5.51 (6.979) | -18.84 (7.051) | 5.48 (7.210)
  48-72 Hours PS (n=81, 89, 74) | 3.23 (9.884) | -6.93 (9.271) | 19.85 (10.568)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 0-24 Hours PS; Test type: Superiority or Other; p = 0.2730, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 0-24 Hours PS; Test type: Superiority or Other; p = 0.1015, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 24-48 Hours PS; Test type: Superiority or Other; p = 0.2438, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 24-48 Hours PS; Test type: Superiority or Other; p = 0.0102, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 48-72 Hours PS; Test type: Superiority or Other; p = 0.2063, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 48-72 Hours PS; Test type: Superiority or Other; p = 0.0387, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

10. Secondary Outcome: Non-opioid Rescue Medication - Paracetamol
Description: The amounts of non-opioid rescue medications, paracetamol, used by the participants during the study, including anti-emetic medications.
Time Frame: 24, 48, 72 hours PS, Discharge (day 3 up to day 7 PS), Week 1, 2, 3, 4 PS,
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Grams (g)
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 150 | 147 | 155
Grams (g)
  24 Hours PS (n=150, 147, 155) | 1.16 (0.098) | 1.21 (0.100) | 1.22 (0.098)
  48 Hours PS (n=150, 147, 154) | 3.23 (0.195) | 3.20 (0.199) | 3.55 (0.195)
  72 Hours PS (n=150, 147,149) | 5.07 (0.294) | 5.08 (0.300) | 5.68 (0.301)
  1st Week PS (n=142, 142, 145) | 10.76 (0.732) | 10.57 (0.739) | 12.63 (0.740)
  2nd Week PS (n=139, 135, 143) | 17.89 (1.711) | 16.79 (1.747) | 19.70 (1.731)
  3rd Week PS (n=131, 124, 134) | 23.56 (2.654) | 22.12 (2.748) | 24.35 (2.695)
  4th Week PS (n=95, 94, 103) | 27.10 (3.313) | 25.62 (3.437) | 25.63 (3.301)
  Till Discharge (n=147, 143, 147) | 5.45 (0.390) | 5.78 (0.399) | 6.05 (0.399)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.5995, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 24 Hours PS; Test type: Superiority or Other; p = 0.9104, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 48 Hours PS; Test type: Superiority or Other; p = 0.2177, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.1770, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.1229, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.1274, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; 1st Week PS; Test type: Superiority or Other; p = 0.0568, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; 1st Week PS; Test type: Superiority or Other; p = 0.0354, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; 2nd Week PS; Test type: Superiority or Other; p = 0.4269, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; 2nd Week PS; Test type: Superiority or Other; p = 0.2058, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; 3rd Week PS; Test type: Superiority or Other; p = 0.8215, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; 3rd Week PS; Test type: Superiority or Other; p = 0.5331, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; 4th Week PS; Test type: Superiority or Other; p = 0.7365, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; 4th Week PS; Test type: Superiority or Other; p = 0.9989, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; Till Discharge; Test type: Superiority or Other; p = 0.2501, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; Till Discharge; Test type: Superiority or Other; p = 0.6021, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

11. Secondary Outcome: Anxiety Before and After Surgery
Description: Participant anxiety reported on Visual Anxiety Scale (VAS), 0 (not at all anxious) to 100 (extremely anxious). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata
Time Frame: Surgery day before first dose and 1 hour after first dose, Day 1, 2, 3, 4, 5 PS and Discharge (day 3 up to day 7 PS)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 150 | 149 | 154
Units on a scale
  Surgery Day (prior to first dose)(n=149, 144, 151) | 31.9 (2.38) | 28.4 (2.45) | 33.3 (2.40)
  Surgery Day (1 hour after dosing)(n=138, 139, 146) | 29.5 (2.39) | 29.7 (2.39) | 30.9 (2.38)
  Day 1 PS (n=150, 149, 154) | 15.6 (1.75) | 16.1 (1.78) | 18.6 (1.77)
  Day 2 PS (n=112, 120, 118) | 12.6 (2.05) | 13.4 (1.98) | 13.8 (2.03)
  Day 3 PS (n=44, 40, 35) | 17.2 (3.17) | 11.2 (2.93) | 13.9 (3.20)
  Day 4 PS (n=17, 20, 15) | 9.0 (3.22) | 4.2 (2.72) | 9.3 (3.51)
  Day 5 PS (n=7, 13, 7) | 11.6 (8.31) | 4.5 (5.39) | 15.1 (8.46)
  Discharge (n=143, 144, 148) | 10.2 (1.50) | 8.3 (1.50) | 8.8 (1.50)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Surgery day (prior to first dose); Test type: Superiority or Other; p = 0.6613, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Surgery day (prior to first dose); Test type: Superiority or Other; p = 0.1311, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Surgery day (1 hour after dosing); Test type: Superiority or Other; p = 0.6574, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Surgery day (1 hour after dosing); Test type: Superiority or Other; p = 0.6949, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 1 PS; Test type: Superiority or Other; p = 0.2008, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 1 PS; Test type: Superiority or Other; p = 0.3022, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.6382, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.8624, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.3858, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.4814, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.9520, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.2315, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.7061, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.2908, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.4782, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.8130, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

12. Secondary Outcome: Non-opioid Rescue Medication - Ibuprofen
Description: The amounts of non-opioid rescue medications, ibuprofen, used by the participants during the study, including anti-emetic medications.
Time Frame: 24, 48, 72 hours PS, Discharge (day 3 up to day 7 PS), Week 1, 2, 3, 4 PS
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Grams (g)
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 150 | 147 | 155
Grams (g)
  24 Hours PS (n=150, 147, 155) | 0.01 (0.014) | 0.03 (0.014) | 0.01 (0.014)
  48 Hours PS (n=150, 147, 154) | 0.08 (0.037) | 0.15 (0.038) | 0.12 (0.038)
  72 Hours PS (n=150, 147, 149) | 0.14 (0.064) | 0.27 (0.065) | 0.24 (0.066)
  1st Week PS (n=142, 142, 145) | 0.51 (0.208) | 0.87 (0.210) | 0.97 (0.211)
  2nd Week PS (n=140, 135, 143) | 1.22 (0.413) | 1.94 (0.423) | 1.88 (0.420)
  3rd Week PS (n=132, 124, 134) | 1.95 (0.665) | 2.99 (0.692) | 2.83 (0.679)
  4th Week PS (n=95, 94, 103) | 2.42 (1.041) | 4.30 (1.080) | 3.84 (1.038)
  Till Discharge (n=147, 143, 147) | 0.18 (0.074) | 0.38 (0.076) | 0.26 (0.076)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.8940, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.5938, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.4306, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.5899, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.2209, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.7145, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; 1st Week PS; Test type: Superiority or Other; p = 0.1022, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; 1st Week PS; Test type: Superiority or Other; p = 0.7243, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; 2nd Week PS; Test type: Superiority or Other; p = 0.2310, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; 2nd Week PS; Test type: Superiority or Other; p = 0.9192, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; 3rd Week PS; Test type: Superiority or Other; p = 0.3214, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; 3rd Week PS; Test type: Superiority or Other; p = 0.8641, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; 4th Week PS; Test type: Superiority or Other; p = 0.3024, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; 4th Week PS; Test type: Superiority or Other; p = 0.7359, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; Till Discharge; Test type: Superiority or Other; p = 0.4303, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; Till Discharge; Test type: Superiority or Other; p = 0.2133, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

13. Secondary Outcome: Percent Change From Baseline in Peak Expiratory Flow
Description: Change from baseline= PEF at x hours minus PEF at baseline; possible values ranged from 0-900 liters/minute (higher values indicated better lung function). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Baseline, every 8 hours (up to 232 hours) PS, and Discharge (Day 3-7 PS flexible)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 116 | 114 | 121
L/min
  Baseline (n=116, 114, 121) | 0 (0) | 0 (0) | 0 (0)
  8 Hours PS (n=84, 79, 83) | -39.25 (3.081) | -35.35 (3.307) | -41.29 (3.242)
  16 Hours PS (n=72, 62, 76) | -37.37 (3.454) | -36.49 (3.764) | -36.48 (3.395)
  24 Hours PS (n=115, 112, 117) | -28.92 (3.084) | -26.53 (3.212) | -29.46 (3.058)
  32 Hours PS (n=104, 105, 106) | -24.53 (3.510) | -25.66 (3.644) | -28.92 (3.632)
  40 Hours PS (n=70, 73, 79) | -24.18 (3.575) | -25.70 (3.663) | -25.07 (3.449)
  48 Hours PS (n=108, 112, 111) | -16.71 (3.203) | -13.62 (3.255) | -21.70 (3.162)
  56 Hours PS (n=78, 85, 82) | -17.11 (3.760) | -15.40 (3.771) | -21.12 (3.726)
  64 Hours PS (n=52, 51, 54) | -15.04 (4.672) | -14.20 (5.028) | -17.18 (4.392)
  72 Hours PS (n=61, 68, 60) | -18.12 (5.270) | -12.97 (4.792) | -20.81 (5.059)
  80 Hours PS (n=30, 24, 24) | -17.23 (7.290) | -3.01 (7.750) | -8.17 (7.443)
  88 Hours PS (n=18, 15, 19) | -10.08 (8.257) | -2.30 (8.818) | -9.71 (6.636)
  96 Hours PS (n=20, 22, 21) | -1.45 (9.063) | 5.26 (8.585) | 2.36 (9.110)
  104 Hours PS (n=9, 12, 12) | -12.79 (10.574) | 0.69 (9.428) | -4.94 (10.210)
  112 Hours PS (n=5, 10, 9) | -15.61 (15.629) | 8.49 (10.863) | -11.61 (10.700)
  120 Hours PS (n=10, 12, 10) | -12.36 (11.386) | -8.14 (10.307) | -6.98 (12.201)
  128 Hours PS (n=4, 9, 7) | -6.72 (13.735) | -4.76 (8.166) | -14.32 (10.711)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; 8 hours PS; Test type: Superiority or Other; p = 0.5682, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; 8 hours PS; Test type: Superiority or Other; p = 0.1005, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; 16 hours PS; Test type: Superiority or Other; p = 0.8261, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; 16 hours PS; Test type: Superiority or Other; p = 0.9981, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.8884, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; 24 hours PS; Test type: Superiority or Other; p = 0.4507, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; 32 hours PS; Test type: Superiority or Other; p = 0.2994, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; 32 hours PS; Test type: Superiority or Other; p = 0.4371, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; 40 hours PS; Test type: Superiority or Other; p = 0.8295, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; 40 hours PS; Test type: Superiority or Other; p = 0.8783, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.2161, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; 48 hours PS; Test type: Superiority or Other; p = 0.0440, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; 56 hours PS; Test type: Superiority or Other; p = 0.3855, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; 56 hours PS; Test type: Superiority or Other; p = 0.2010, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; 64 hours PS; Test type: Superiority or Other; p = 0.7104, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; 64 hours PS; Test type: Superiority or Other; p = 0.6107, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 17: Comparison: Pregabalin 150mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.6705, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; 72 hours PS; Test type: Superiority or Other; p = 0.2083, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 19: Comparison: Pregabalin 150mg vs Placebo; 80 hours PS; Test type: Superiority or Other; p = 0.3234, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 20: Comparison: Pregabalin 300 mg vs Placebo; 80 hours PS; Test type: Superiority or Other; p = 0.5938, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 21: Comparison: Pregabalin 150mg vs Placebo; 88 hours PS; Test type: Superiority or Other; p = 0.9711, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 22: Comparison: Pregabalin 300 mg vs Placebo; 88 hours PS; Test type: Superiority or Other; p = 0.4869, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 23: Comparison: Pregabalin 150mg vs Placebo; 96 hours PS; Test type: Superiority or Other; p = 0.7439, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 24: Comparison: Pregabalin 300 mg vs Placebo; 96 hours PS; Test type: Superiority or Other; p = 0.8045, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 25: Comparison: Pregabalin 150mg vs Placebo; 104 hours PS; Test type: Superiority or Other; p = 0.5925, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 26: Comparison: Pregabalin 300 mg vs Placebo; 104 hours PS; Test type: Superiority or Other; p = 0.6830, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 27: Comparison: Pregabalin 150mg vs Placebo; 112 hours PS; Test type: Superiority or Other; p = 0.8266, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 28: Comparison: Pregabalin 300 mg vs Placebo; 112 hours PS; Test type: Superiority or Other; p = 0.1929, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 29: Comparison: Pregabalin 150mg vs Placebo; 120 hours PS; Test type: Superiority or Other; p = 0.7071, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 30: Comparison: Pregabalin 300 mg vs Placebo; 120 hours PS; Test type: Superiority or Other; p = 0.9367, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 31: Comparison: Pregabalin 150mg vs Placebo; 128 hours PS; Test type: Superiority or Other; p = 0.6046, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 32: Comparison: Pregabalin 300 mg vs Placebo; 128 hours PS; Test type: Superiority or Other; p = 0.5119, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

14. Secondary Outcome: Timed Up-and-Go (TUG)
Description: Functional mobility test performed once a day at 24 hour intervals from surgery after the pain with movement assessment. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Day 1, 2, 3, 4, 5 PS and Discharge (day 3 up to day 7 PS)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 130 | 134 | 134
Seconds
  Day 1 PS (n=85, 85, 93) | 39.77 (2.558) | 42.79 (2.769) | 38.54 (2.611)
  Day 2 PS (n=107, 105, 105) | 31.82 (1.776) | 33.06 (1.878) | 29.25 (1.845)
  Day 3 PS (n=43, 35, 31) | 34.07 (2.779) | 33.48 (2.781) | 31.38 (2.960)
  Day 4 PS (n=16, 18, 13) | 42.26 (4.591) | 37.31 (4.065) | 40.43 (5.275)
  Day 5 PS (n=7, 10, 7) | 31.27 (5.295) | 23.06 (3.704) | 32.18 (5.326)
  Discharge (n=130, 134, 134) | 28.11 (1.604) | 30.05 (1.569) | 26.40 (1.582)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 1 PS; Test type: Superiority or Other; p = 0.6966, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 1 PS; Test type: Superiority or Other; p = 0.1808, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.2616, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.1014, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.4401, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.5615, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.7615, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.6204, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.8766, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.1717, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.4065, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0746, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

15. Secondary Outcome: Average Daily Pain
Description: Post-discharge average pain as measured in daily participant diaries NRS an 11 point Likert scale ranged from 0 (no pain) to 10 (worst pain). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Day 2, 3, 4, 5, 6, 7, PS; week 2, 3, 4 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 134 | 131 | 139
Units on a scale
  Day 2 PS (n=29, 21, 25) | 3.9 (0.48) | 4.3 (0.55) | 3.1 (0.59)
  Day 3 PS (n=97, 94, 98) | 3.0 (0.22) | 3.2 (0.23) | 2.8 (0.23)
  Day 4 PS (n=126, 114, 125) | 2.7 (0.19) | 2.9 (0.21) | 2.8 (0.20)
  Day 5 PS (n=133, 117, 133) | 2.5 (0.18) | 2.6 (0.20) | 2.6 (0.19)
  Day 6 PS (n=133, 125, 138) | 2.3 (0.18) | 2.5 (0.19) | 2.4 (0.18)
  Day 7 PS (n=132, 130, 135) | 2.1 (0.17) | 2.3 (0.17) | 2.2 (0.17)
  2nd Week PS (Average) (n=134, 131, 139) | 1.7 (0.14) | 2.0 (0.14) | 1.7 (0.14)
  3rd Week PS (Average) (n=114, 110, 114) | 1.3 (0.15) | 1.7 (0.15) | 1.3 (0.16)
  4th Week PS (Average) (n=87, 87, 82) | 1.2 (0.18) | 1.6 (0.19) | 1.2 (0.20)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.2201, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.0606, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.5303, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.2227, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.8237, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.7476, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.6882, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.9689, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Day 6 PS; Test type: Superiority or Other; p = 0.5010, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Day 6 PS; Test type: Superiority or Other; p = 0.9143, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Day 7 PS; Test type: Superiority or Other; p = 0.7381, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Day 7 PS; Test type: Superiority or Other; p = 0.5336, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; 2nd Week PS (Average); Test type: Superiority or Other; p = 0.6479, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; 2nd Week PS (Average); Test type: Superiority or Other; p = 0.1133, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; 3rd Week PS (Average); Test type: Superiority or Other; p = 0.7637, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; 3rd Week PS (Average); Test type: Superiority or Other; p = 0.1056, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 17: Comparison: Pregabalin 150mg vs Placebo; 4th Week PS (Average); Test type: Superiority or Other; p = 0.8079, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; 4th Week PS (Average); Test type: Superiority or Other; p = 0.0917, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

16. Secondary Outcome: Worst Daily Pain
Description: Post-discharge worst pain as measured in daily participant diaries NRS an 11 point Likert scale that ranged from 0 (no pain) to 10 (pain as bad as you can imagine). LS Means from ANOVA model with terms of treatment, pooled center, salpingo-oophorectomy strata and baseline worst pain score.
Time Frame: Discharge (day 3 up to day 7 PS), Day 7, 14, 28 PS
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 141 | 143 | 143
Units on a scale
  Discharge (n=140, 143, 138) | 4.3 (0.22) | 4.4 (0.22) | 4.2 (0.22)
  Day 7 (n=123, 121, 125) | 3.2 (0.24) | 3.4 (0.24) | 3.5 (0.23)
  Day 14 (n=129, 125, 130) | 1.8 (0.19) | 2.4 (0.19) | 2.5 (0.19)
  Day 28 (n=141, 142, 143) | 1.2 (0.15) | 1.7 (0.15) | 1.4 (0.15)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.7511, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.6742, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.3808, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.7021, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0045, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.7916, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.3682, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.1419, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

17. Secondary Outcome: Sleep Interference
Description: Sleep interference post surgery measured daily in participant diaries; NRS of how pain interfered with sleep during the last 24 hours, ranged from 0 (does not interfere) to 10 (completely interferes). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Daily post hospital discharge ( Day 2-7 PS), Week 2, 3, 4 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 134 | 131 | 139
Units on a scale
  Day 2 PS (n=21, 18, 20) | 2.4 (0.65) | 3.6 (0.67) | 3.2 (0.77)
  Day 3 PS (n=88, 89, 87) | 2.6 (0.32) | 2.3 (0.33) | 2.6 (0.33)
  Day 4 PS (n=122, 111, 119) | 2.3 (0.24) | 2.5 (0.27) | 2.5 (0.26)
  Day 5 PS (n=133, 117, 132) | 2.1 (0.22) | 2.2 (0.24) | 2.5 (0.22)
  Day 6 PS (n=133, 127, 138) | 1.7 (0.22) | 1.9 (0.23) | 2.1 (0.22)
  Day 7 PS (n=132, 131, 138) | 1.7 (0.22) | 2.0 (0.22) | 2.1 (0.22)
  2nd Week PS (Average) (n=134, 131, 139) | 1.3 (0.16) | 1.7 (0.17) | 1.5 (0.16)
  3rd Week PS (Average) (n=115, 112, 113) | 1.0 (0.16) | 1.3 (0.16) | 1.0 (0.17)
  4th Week PS (Average) (n=87, 87, 81) | 1.0 (0.21) | 1.4 (0.21) | 0.9 (0.22)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.3323, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.5662, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.9538, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.4592, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.4793, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.8517, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.1829, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.3544, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Day 6 PS; Test type: Superiority or Other; p = 0.1718, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Day 6 PS; Test type: Superiority or Other; p = 0.5078, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Day 7 PS; Test type: Superiority or Other; p = 0.2443, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Day 7 PS; Test type: Superiority or Other; p = 0.8296, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; 2nd Week PS (Average); Test type: Superiority or Other; p = 0.3243, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; 2nd Week PS (Average); Test type: Superiority or Other; p = 0.3755, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; 3rd Week PS (Average); Test type: Superiority or Other; p = 0.9584, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; 3rd Week PS (Average); Test type: Superiority or Other; p = 0.1187, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 17: Comparison: Pregabalin 150mg vs Placebo; 4th Week PS (Average); Test type: Superiority or Other; p = 0.7915, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; 4th Week PS (Average); Test type: Superiority or Other; p = 0.0703, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

18. Secondary Outcome: Brief Pain Inventory-Short Form (m-BPI-sf): Pain Interference Index Scores
Description: m-BPI-sf: participant-rated 11 point Likert rating scale ranging from 0 (does not interfere) to 10 (completely interferes) with functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Baseline, Discharge (day 3 up to day 7 PS), Day 7, 14, 28 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 149 | 147 | 154
Units on a scale
  Baseline (n=149, 147, 154) | 0 (0) | 0 (0) | 0 (0)
  Discharge (n=133, 131, 130) | 2.57 (0.194) | 2.62 (0.198) | 2.90 (0.200)
  Day 7 (n=121, 119, 123) | 1.96 (0.201) | 2.09 (0.206) | 2.52 (0.198)
  Day 28 (n=140, 141, 142) | 0.85 (0.122) | 1.01 (0.122) | 1.07 (0.123)
  Day 14 (n=129, 123, 126) | 1.20 (0.148) | 1.41 (0.152) | 1.68 (0.152)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Discharge;; Test type: Superiority or Other; p = 0.1975, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Discharge;; Test type: Superiority or Other; p = 0.2784, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0271, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0881, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0159, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.1870, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.1752, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.6923, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

19. Other Pre Specified Outcome: Percentage of Participants With Wound Healing Complications - Discharge
Description: Pre-specified adverse events of wound healing complications based on Center for Disease Control and Prevention, 1999, guidelines for prevention of surgical site infection (SSI) wound healing complications included: superficial incisional SSI, deep incisional SSI, organ/space SSI or non-infections wound healing complication.
Time Frame: Discharge (day 3 up to day 7 PS)
Population: Safety population all participants who were administered at least one dose of double blind medication, and for whom at least one post-baseline safety evaluation was obtained were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 161 | 166 | 167
Percentage of participants
  Superficial Incision SSI | 3.1 | 1.2 | 0.6
  Deep Incision SSI | 0 | 0 | 0
  Organ/space SSI | 0 | 0 | 0
  Non-infectious Wound Healing | 0 | 1.2 | 0

20. Other Pre Specified Outcome: Percentage of Participants With Wound Healing Complications - Day 7 PS
Description: as for outcome 19
Time Frame: Day 7 PS
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 161 | 166 | 167
Percentage of participants
  Superficial Incision SSI | 1.9 | 2.5 | 0.6
  Deep Incision SSI | 0.6 | 0 | 0
  Organ/space SSI | 0 | 0 | 0
  Non-infectious Wound Healing | 3.8 | 1.9 | 0.6

21. Secondary Outcome: Brief Pain Inventory-Short Form (m-BPI-sf): Pain Severity Index Scores
Description: m-BPI-sf: participant rated 11-point Likert rating scale ranging from 0 (no pain) to 10 (worst pain possible). Pain severity index is the mean of item scores 2, 3, and 4 (pain right now, worst pain, and average pain level).
  LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Baseline, Discharge (day 3 up to day 7 PS), Day 7, 14, 28 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 149 | 147 | 155
Units on a scale
  Baseline (n=149, 147, 155) | 0 (0) | 0 (0) | 0 (0)
  Discharge (n=140, 141, 138) | 2.62 (0.137) | 2.60 (0.137) | 2.53 (0.141)
  Day 7 (n=122, 121, 125) | 2.05 (0.172) | 2.16 (0.177) | 2.20 (0.169)
  Day 14 (n=129, 124, 130) | 1.19 (0.137) | 1.63 (0.142) | 1.61 (0.138)
  Day 28 (n=141, 142, 143) | 0.79 (0.110) | 0.98 (0.110) | 0.83 (0.110)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.6295, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.6890, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.5094, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.8741, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0214, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.9366, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.7833, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.2983, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

22. Other Pre Specified Outcome: Percentage of Participants With Wound Healing Complications - Day 14 PS
Description: as for outcome 19
Time Frame: Day 14 PS
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 161 | 166 | 167
Percentage of participants
  Superficial Incision SSI | 5.0 | 2.5 | 2.4
  Deep Incision SSI | 0.6 | 0 | 0
  Organ/space SSI | 0.6 | 0 | 0
  Non-infectious Wound Healing | 4.4 | 2.5 | 0.6

23. Other Pre Specified Outcome: Percentage of Participants With Wound Healing Complications - Day 28 PS
Description: as for outcome 19
Time Frame: Day 28 PS
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 161 | 166 | 167
Percentage of participants
  Superficial Incision SSI | 1.9 | 1.9 | 1.2
  Deep Incision SSI | 0 | 0 | 0
  Organ/space SSI | 0 | 0 | 0.6
  Non-infectious Wound Healing | 2.5 | 2.5 | 0

24. Secondary Outcome: Participant Satisfaction With Study Medication - Surgery Day
Description: Participant satisfaction with study medication using the Global Evaluation of Study Medication questionaire. Participants overall impression (global evaluation) of the study medication was recorded by the participant by answering the following question: How would you rate the study medication you received for pain? Excellent 4; Good 3; Fair 2; Poor 1.
Time Frame: Day 1
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 40
Percentage of participants
  Excellent | 14.3 | 3.1 | 20.0
  Good | 42.9 | 62.5 | 35.0
  Fair | 39.3 | 31.3 | 30.0
  Poor | 3.6 | 3.1 | 15.0
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Surgery Day; Test type: Superiority or Other; p = 0.6861, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Surgery Day; Test type: Superiority or Other; p = 0.9905, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

25. Secondary Outcome: Participant Satisfaction With Study Medication - Day 1 PS
Description: as for outcome 24
Time Frame: Day 1 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 150 | 148 | 154
Percentage of participants
  Excellent | 13.3 | 17.6 | 16.2
  Good | 56.0 | 47.3 | 45.5
  Fair | 26.7 | 29.1 | 30.5
  Poor | 4.0 | 6.1 | 7.8
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 1 PS; Test type: Superiority or Other; p = 0.4264, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 1 PS; Test type: Superiority or Other; p = 0.3045, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

26. Secondary Outcome: Participant Satisfaction With Study Medication - Day 2 PS
Description: as for outcome 24
Time Frame: Day 2 PS
Population: mITT; N=number of evaluable participants analyzed;
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 114 | 119 | 117
Percentage of participants
  Excellent | 21.9 | 17.6 | 16.2
  Good | 49.1 | 54.6 | 47.0
  Fair | 25.4 | 21.8 | 29.1
  Poor | 3.5 | 5.9 | 7.7
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.0714, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 2 PS; Test type: Superiority or Other; p = 0.4455, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

27. Secondary Outcome: Participant Satisfaction With Study Medication - Day 3 PS
Description: as for outcome 24
Time Frame: Day 3 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 44 | 40 | 34
Percentage of participants
  Excellent | 15.9 | 17.5 | 17.6
  Good | 52.3 | 47.5 | 50.0
  Fair | 31.8 | 30.0 | 29.4
  Poor | 0 | 5.0 | 2.9
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.7418, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 3 PS; Test type: Superiority or Other; p = 0.5154, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

28. Secondary Outcome: Participant Satisfaction With Study Medication - Day 4 PS
Description: as for outcome 24
Time Frame: Day 4 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 17 | 19 | 14
Percentage of participants
  Excellent | 17.6 | 5.3 | 14.3
  Good | 52.9 | 57.9 | 42.9
  Fair | 29.4 | 31.6 | 28.6
  Poor | 0 | 5.3 | 14.3
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.6715, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 4 PS; Test type: Superiority or Other; p = 0.9013, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

29. Secondary Outcome: Participant Satisfaction With Study Medication - Day 5 PS
Description: as for outcome 24
Time Frame: Day 5 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 7 | 13 | 7
Percentage of participants
  Excellent | 0 | 7.7 | 14.3
  Good | 71.4 | 53.8 | 42.9
  Fair | 28.6 | 38.5 | 28.6
  Poor | 0 | 0 | 14.3
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 0.9126, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 5 PS; Test type: Superiority or Other; p = 1.0000, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

30. Secondary Outcome: Participant Satisfaction With Study Medication - Discharge
Description: as for outcome 24
Time Frame: Discharge (day 3 up to day 7 PS)
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 142 | 145 | 148
Percentage of participants
  Excellent | 29.6 | 26.2 | 26.4
  Good | 48.6 | 51.0 | 39.9
  Fair | 16.9 | 17.9 | 25.0
  Poor | 4.9 | 4.8 | 8.8
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1233, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1666, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

31. Secondary Outcome: Participant Satisfaction With Study Medication - Day 7 PS
Description: as for outcome 24
Time Frame: Day 7 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 123 | 122 | 127
Percentage of participants
  Excellent | 36.6 | 36.9 | 25.2
  Good | 38.2 | 37.7 | 39.4
  Fair | 15.4 | 17.2 | 26.0
  Poor | 9.8 | 8.2 | 9.4
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0361, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0797, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

32. Secondary Outcome: Participant Satisfaction With Study Medication - Day 14 PS
Description: as for outcome 24
Time Frame: Day 14 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 130 | 126 | 131
Percentage of participants
  Excellent | 40.0 | 42.9 | 31.3
  Good | 42.3 | 37.3 | 33.6
  Fair | 11.5 | 16.7 | 24.4
  Poor | 6.2 | 3.2 | 10.7
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0206, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

33. Other Pre Specified Outcome: Percentage of Participants With Wound Healing Complications - End of Treatment
Description: as for outcome 19
Time Frame: Day 1 up to Day 28 PS
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 161 | 166 | 167
Percentage of participants
  Superficial Incision SSI | 0 | 1.2 | 0
  Deep Incision SSI | 0 | 0 | 0
  Organ/space SSI | 0 | 0 | 0
  Non-infectious Wound Healing | 0 | 0 | 0

34. Other Pre Specified Outcome: Incision Length Correlated With Worst Pain
Description: Incision length (cm) correlated with worst pain. Worst pain ranged from 0 (no pain) to 10 (worst pain imaginable). LS Means adjusted for treatment, pooled center, salpingo-oophorectomy strata.
Time Frame: Day 1
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: Centimeter (cm)
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 151 | 149 | 156
Centimeter (cm) | 7.1074 (0.2010) | 7.2324 (0.1966) | 7.4437 (0.1977)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Pregabalin 300 mg vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.3506, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

35. Secondary Outcome: Participant Satisfaction With Study Medication - Day 28 PS
Description: as for outcome 24
Time Frame: Day 28 PS
Population: mITT; N=number of evaluable participants analyzed
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 139 | 142 | 143
Percentage of participants
  Excellent | 42.4 | 40.1 | 34.3
  Good | 41.7 | 34.5 | 35.0
  Fair | 9.4 | 16.2 | 23.8
  Poor | 6.5 | 9.2 | 7.0
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.0287, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.2270, Cochran-Mantel-Haenszel; CMH test adjusted for pooled centers and salpingo-oophorectomy strata

36. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Satisfaction With Current Pain Medication
Description: Satisfaction with current pain medication ranged from 0 (worst possible response) to100 (best possible response). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Discharge (day 3 up to day 7 PS), Day 28 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 138 | 137 | 139
Units on a scale
  Medication Subscale/Discharge (n=138, 137, 139) | 79.43 (1.717) | 78.45 (1.747) | 76.71 (1.776)
  Medication Subscale/Day 28 (n=133, 134, 137) | 82.52 (1.619) | 80.16 (1.601) | 78.26 (1.615)
  Characteristic Subscale/Discharge (n=138,136,138) | 82.15 (1.565) | 81.88 (1.597) | 79.58 (1.623)
  Characteristic Subscale/Day 28 (n=133, 133, 137) | 84.82 (1.448) | 83.16 (1.438) | 81.69 (1.445)
  Efficacy Subscale/Discharge (n=138, 137, 139) | 76.68 (2.264) | 75.04 (2.304) | 73.77 (2.342)
  Efficacy Subscale/Day 28 (n=133, 134, 136) | 80.20 (2.161) | 76.92 (2.138) | 74.82 (2.166)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Medication Subscale at Discharge; Test type: Superiority or Other; p = 0.1872, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Medication Subscale at Discharge; Test type: Superiority or Other; p = 0.3994, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Medication Subscale at Day 28; Test type: Superiority or Other; p = 0.0422, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Medication Subscale at Day 28; Test type: Superiority or Other; p = 0.3647, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Characteristics at Discharge; Test type: Superiority or Other; p = 0.1729, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Characteristics at Discharge; Test type: Superiority or Other; p = 0.2234, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Characteristics at Day 28; Test type: Superiority or Other; p = 0.0950, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Characteristics at Day 28; Test type: Superiority or Other; p = 0.4345, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Efficacy at Discharge; Test type: Superiority or Other; p = 0.2840, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Efficacy at Discharge; Test type: Superiority or Other; p = 0.6404, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Efficacy at Day 28; Test type: Superiority or Other; p = 0.0550, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Efficacy at Day 28; Test type: Superiority or Other; p = 0.4531, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

37. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Impact of Current Pain Medication
Description: Impact of current pain medication response scale: 0 (worst possible response) to 100 (best possible response). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Discharge (day 3 up to day 7 PS), Day 28 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 139 | 141 | 141
Units on a scale
  Discharge (n=139, 141, 140) | 72.73 (2.080) | 66.28 (2.099) | 72.82 (2.159)
  Day 28 (n=133, 135, 141) | 76.41 (2.180) | 69.53 (2.181) | 69.05 (2.156)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.9712, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0112, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.0090, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.8650, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

38. Secondary Outcome: Quality of Life Using EuroQol (EQ-5D) Health State Profile
Description: Participant rated questionnaire assessed current health for 6 domains: mobility/self-care/ usual activities/pain/discomfort/anxiety and depression. Scoring developed by EuroQol Group assigned a utility value for each domain in the profile. Scores ranged from 1 better health (no problems) to 3 worst health (eg, "confined to bed"). Score transformed and resulted in a total score range -0.594 to 1.000; higher score=better health state. Health profile scores estimated using Dolan computational algorithms 1997 and 2001. LS Means adjusted for treatment/pooled center/salpingo-oophorectomy strata.
Time Frame: Discharge (day 3 up to day 7 PS) and day 28 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 140 | 143 | 142
Units on a scale
  EQ-5D 1997, Discharge (n=138, 141, 138) | 0.57 (0.021) | 0.61 (0.021) | 0.58 (0.022)
  EQ-5D 1997, Day 28 (n=140, 143, 142) | 0.81 (0.014) | 0.78 (0.014) | 0.78 (0.014)
  EQ-5D 2001, Discharge (n=138, 141, 138) | 0.59 (0.018) | 0.62 (0.018) | 0.60 (0.019)
  EQ-5D 2001, Day 28 (n=140, 143, 142) | 0.81 (0.014) | 0.78 (0.014) | 0.78 (0.014)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; EQ-5D 1997 Discharge; Test type: Superiority or Other; p = 0.8914, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; EQ-5D 1997 Discharge; Test type: Superiority or Other; p = 0.2214, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; EQ-5D 1997 Day 28; Test type: Superiority or Other; p = 0.1008, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; EQ-5D 1997 Day 28; Test type: Superiority or Other; p = 0.9135, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; EQ-5D 2001 Discharge; Test type: Superiority or Other; p = 0.5609, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; EQ-5D 2001 Discharge; Test type: Superiority or Other; p = 0.4047, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; EQ-5D 2001 Day 28; Test type: Superiority or Other; p = 0.1663, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; EQ-5D 2001 Day 28; Test type: Superiority or Other; p = 0.8364, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

39. Secondary Outcome: Time to Meet Hospital Discharge Criteria
Description: Mean time from end of surgery to meet protocol defined hospital discharge criteria: participant no longer received parental opioids, was able to dress and mobilize without assistance, and had normal intake of food and fluids.
Time Frame: Day 1 up to Day 7 PS
Population: mITT
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 151 | 149 | 156
Hours | 57.670 (2.829) | 60.751 (2.678) | 58.745 (2.786)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Kaplan-Meier method was used for survival distribution estimation;; Test type: Superiority or Other; p = 0.7218, Log Rank
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Kaplan-Meier method was used for survival distribution estimation;; Test type: Superiority or Other; p = 0.4425, Log Rank

40. Secondary Outcome: Time to Actual Discharge
Description: Mean time from end of surgery to actual hospital discharge. Participant was expected to remain at the hospital for a minimum of 2 days following surgery.
Time Frame: Day 1 up to Day 7 PS
Population: mITT
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 151 | 149 | 156
Hours | 79.339 (2.547) | 85.221 (3.935) | 78.740 (2.441)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Kaplan-Meier method was used for survival distribution estimation;; Test type: Superiority or Other; p = 0.7889, Log Rank
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Kaplan-Meier method was used for survival distribution estimation;; Test type: Superiority or Other; p = 0.1565, Log Rank

41. Other Pre Specified Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: Pain characteristics in participants who reported pain (mBPI-sf, NPSI); NPSI a participant rated questionnaire to evaluate different symptoms of neuropathic pain, burning spontaneous pain, pressing spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia at discharge. NPSI Total Score ranged from 0 to 0.5; NPSI subscales pain ranged from 0 (no pain) to 10 (worst pain). LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Discharge (day 3 up to day 7 PS)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 139 | 145 | 143
Units on a scale
  Total subscale(n=132, 131, 136) | 0.073 (0.0057) | 0.070 (0.0057) | 0.076 (0.0058)
  Burning Spontaneous subscale (n=139, 145, 143) | 1.86 (0.235) | 1.80 (0.231) | 1.75 (0.235)
  Pressing Spontaneous subscale (n=139, 145, 143) | 1.74 (0.166) | 1.60 (0.164) | 1.57 (0.168)
  Paroxysmal pain subscale (n=138, 140, 143) | 1.08 (0.155) | 0.95 (0.154) | 1.18 (0.156)
  Evoked Pain subscale (n=134, 135, 142) | 2.14 (0.177) | 2.27 (0.177) | 2.27 (0.175)
  Paresthesia/dysesthesia (n=136, 140, 141) | 0.46 (0.129) | 0.67 (0.127) | 0.91 (0.128)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Total subscale; Test type: Superiority or Other; p = 0.6211, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Total subscale; Test type: Superiority or Other; p = 0.3687, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Burning Spontaneous subscale; Test type: Superiority or Other; p = 0.7078, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Burning Spontaneous subscale; Test type: Superiority or Other; p = 0.8696, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Pressing Spontaneous subscale; Test type: Superiority or Other; p = 0.4320, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Pressing Spontaneous subscale; Test type: Superiority or Other; p = 0.8843, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Paroxysmal pain subscale; Test type: Superiority or Other; p = 0.6215, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Paroxysmal pain subscale; Test type: Superiority or Other; p = 0.2722, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Evoked Pain subscale; Test type: Superiority or Other; p = 0.5500, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Evoked Pain subscale; Test type: Superiority or Other; p = 0.9942, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Paresthesia/dysesthesia; Test type: Superiority or Other; p = 0.0075, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Paresthesia/dysesthesia; Test type: Superiority or Other; p = 0.1464, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

42. Secondary Outcome: Incidence of Chronic Post-operative Pain
Description: Chronic post-operative pain as a result of abdominal hysterectomy as reported by participants on PS questionaire of pain within last 24 hours in area affected by surgery.
Time Frame: 3 and 6 Months PS
Population: mITT; n = number of evaluable participants analyzed for the given time point; N=number of evaluable participants analyzed. Participants reported as no chronic pain in the 3 month visit were carried over to the missing data at 6 month visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 138 | 127 | 141
Percentage of participants
  Months 3 PS (n =136, 127, 138) | 12.5 | 17.3 | 10.1
  Months 6 PS (n =138, 127, 141) | 6.5 | 6.3 | 4.3
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Incidence of chronic PS pain at Month 3 PS; Test type: Superiority or Other; p = 0.9877, Cochran-Mantel-Haenszel; p-values are derived from CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Incidence of chronic PS pain at Month 3 PS; Test type: Superiority or Other; p = 0.1334, Cochran-Mantel-Haenszel; p-values are derived from CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Incidence of chronic PS pain at Month 6 PS; Test type: Superiority or Other; p = 0.3566, Cochran-Mantel-Haenszel; p-values are derived from CMH test adjusted for pooled centers and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Incidence of chronic PS pain at Month 6 PS; Test type: Superiority or Other; p = 0.6262, Cochran-Mantel-Haenszel; p-values are derived from CMH test adjusted for pooled centers and salpingo-oophorectomy strata

43. Secondary Outcome: Total Clinically Meaningful Event (CME) Score
Description: Total CME score calculated by summing the number of Clinically Meaningful Events (CMEs) across symptoms. CME for each symptom will be defined using the Opioid-Related Symptom Distress Scale (OR-SDS) a participant rated scale of symptoms within the last 24 hours. Total CME score could range from 0 to 9. LS Means adjusted for treatment, pooled center and salpingo-oophorectomy strata.
Time Frame: Surgery Day, Day 1, 2, 3, 4, 5 PS, Discharge (day 3 up to day 7 PS), Day 7, 14, 28 PS
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Number analyzed (Participants) | 148 | 147 | 154
Units on a scale
  Surgery Day (n=26, 25, 32) | 0.9 (0.29) | 0.8 (0.30) | 0.9 (0.26)
  Day 1 PS (n=148, 147, 154) | 1.1 (0.13) | 1.1 (0.13) | 1.2 (0.13)
  Day 2 PS (n=108, 116, 114) | 0.6 (0.12) | 0.6 (0.12) | 0.7 (0.12)
  Day 3 PS (n=38, 36, 32) | 0.5 (0.19) | 0.7 (0.17) | 0.3 (0.19)
  Day 4 PS (n=14, 16, 11) | 0.0 (0.19) | 0.4 (0.15) | 0.3 (0.22)
  Day 5 PS (n=5, 9, 6) | 0.4 (0.19) | 0.1 (0.13) | 0.3 (0.18)
  Discharge (n=133, 132, 133) | 0.4 (0.09) | 0.4 (0.09) | 0.3 (0.09)
  Day 7 PS (n=119, 117, 120) | 0.2 (0.06) | 0.4 (0.06) | 0.2 (0.06)
  Day 14 PS (n=119, 116, 124) | 0.1 (0.06) | 0.2 (0.06) | 0.1 (0.06)
  Day 28 PS (n=129, 135, 136) | 0.0 (0.06) | 0.2 (0.06) | 0.2 (0.06)
Statistical Analysis 1: Comparison: Pregabalin 150mg vs Placebo; Surgery day;; Test type: Superiority or Other; p = 0.9463, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Placebo; Surgery day;; Test type: Superiority or Other; p = 0.7347, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 3: Comparison: Pregabalin 150mg vs Placebo; Day 1 PS;; Test type: Superiority or Other; p = 0.4132, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 4: Comparison: Pregabalin 300 mg vs Placebo; Day 1 PS;; Test type: Superiority or Other; p = 0.4929, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 5: Comparison: Pregabalin 150mg vs Placebo; Day 2 PS;; Test type: Superiority or Other; p = 0.6003, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 6: Comparison: Pregabalin 300 mg vs Placebo; Day 2 PS;; Test type: Superiority or Other; p = 0.9343, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 7: Comparison: Pregabalin 150mg vs Placebo; Day 3 PS;; Test type: Superiority or Other; p = 0.3838, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 8: Comparison: Pregabalin 300 mg vs Placebo; Day 3 PS;; Test type: Superiority or Other; p = 0.1351, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 9: Comparison: Pregabalin 150mg vs Placebo; Day 4 PS;; Test type: Superiority or Other; p = 0.3343, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 10: Comparison: Pregabalin 300 mg vs Placebo; Day 4 PS;; Test type: Superiority or Other; p = 0.7948, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 11: Comparison: Pregabalin 150mg vs Placebo; Day 5 PS;; Test type: Superiority or Other; p = 0.8090, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 12: Comparison: Pregabalin 300 mg vs Placebo; Day 5 PS;; Test type: Superiority or Other; p = 0.4035, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 13: Comparison: Pregabalin 150mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.6009, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 14: Comparison: Pregabalin 300 mg vs Placebo; Discharge; Test type: Superiority or Other; p = 0.7597, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 15: Comparison: Pregabalin 150mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.7804, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 16: Comparison: Pregabalin 300 mg vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0463, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 17: Comparison: Pregabalin 150mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.4951, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 18: Comparison: Pregabalin 300 mg vs Placebo; Day 14; Test type: Superiority or Other; p = 0.3030, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 19: Comparison: Pregabalin 150mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.0104, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata
Statistical Analysis 20: Comparison: Pregabalin 300 mg vs Placebo; Day 28; Test type: Superiority or Other; p = 0.6978, ANOVA; LS Means from ANOVA model with terms of treatment, pooled center and salpingo-oophorectomy strata

ADVERSE EVENTS:
Arm/Group | Pregabalin 150mg | Pregabalin 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/161 | 11/166 | 15/167
Other Adverse Events (participants affected / at risk) | 125/161 | 128/166 | 124/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 150mg (N=161) | Pregabalin 300 mg (N=166) | Placebo (N=167)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Incision site infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 2 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ureteric injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 150mg (N=161) | Pregabalin 300 mg (N=166) | Placebo (N=167)
Anaemia (Blood and lymphatic system disorders) | 9 | 5 | 5
Tachycardia (Cardiac disorders) | 4 | 6 | 3
Vision blurred (Eye disorders) | 2 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 6 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 4 | 10
Constipation (Gastrointestinal disorders) | 46 | 49 | 45
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 5 | 6 | 6
Flatulence (Gastrointestinal disorders) | 16 | 10 | 13
Nausea (Gastrointestinal disorders) | 67 | 60 | 76
Retching (Gastrointestinal disorders) | 0 | 6 | 4
Vomiting (Gastrointestinal disorders) | 33 | 20 | 30
Chills (General disorders) | 1 | 2 | 4
Fatigue (General disorders) | 38 | 46 | 34
Oedema peripheral (General disorders) | 4 | 1 | 1
Pain (General disorders) | 4 | 3 | 3
Pyrexia (General disorders) | 31 | 29 | 24
Urinary tract infection (Infections and infestations) | 13 | 12 | 8
Wound infection (Infections and infestations) | 5 | 5 | 3
Procedural pain (Injury, poisoning and procedural complications) | 2 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 4
Disturbance in attention (Nervous system disorders) | 24 | 30 | 23
Dizziness (Nervous system disorders) | 51 | 52 | 37
Headache (Nervous system disorders) | 27 | 23 | 19
Hypoaesthesia (Nervous system disorders) | 0 | 4 | 4
Migraine (Nervous system disorders) | 2 | 4 | 2
Paraesthesia (Nervous system disorders) | 4 | 0 | 2
Somnolence (Nervous system disorders) | 39 | 39 | 36
Confusional state (Psychiatric disorders) | 12 | 12 | 9
Insomnia (Psychiatric disorders) | 9 | 9 | 10
Dysuria (Renal and urinary disorders) | 14 | 22 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 22 | 26
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Haematoma (Vascular disorders) | 6 | 6 | 2
Hypertension (Vascular disorders) | 3 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other